CLINICAL TRIAL: NCT05178927
Title: UFPTI 2105-BR05: Improving Breast Radiotherapy Setup and Delivery Using Mixed-Reality Visualization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB202101449
Record Dates: First submitted 2021-10-11; First posted 2022-01-05 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care-Group 1 (Sham Comparator): During treatments 1-5, radiation therapists will position the participant for treatment using the standard of care method.
  During treatments 6-10, radiation therapists will use the hologram the investigators created to initially position the participant for treatment. The participant's final position will be obtained using a standard of care method.
  Interventions: Device: HoloLens v2
- Mixed-reality guided patient setup-Group 2 (Experimental): During treatments 1-5, radiation therapists will use the hologram the investigators created to initially position the participant for treatment. The participant's final position will be obtained using a standard of care method.
  During treatments 6-10, radiation therapists will position the participant for treatment using the standard of care method.
  Interventions: Device: HoloLens v2

INTERVENTIONS:
Device: HoloLens v2 — The HoloLens v2 will be used to access the participant's hologram & set the participant up for treatment. Standard of care methods will be utilized to confirm treatment set-up.

SUMMARY:
The purpose of this study is to compare the accuracy, set-up time, and amount of image-guided radiotherapy (IGRT - a system that helps line up the radiation beam with the tumor for treatment) needed when mixed-reality guided radiotherapy is used for treatment set-up.

ELIGIBILITY:
Inclusion Criteria:

* Targets adult patients who are planning to undergo photon or proton radiation therapy at UFHPTI for treatment of the breast or chest wall. As this type of treatment is rare in men, the study will focus on female patients only.

Exclusion Criteria:

* Male subjects

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As this type of treatment is rare in men, the study will focus on female patients only.
Enrollment: 27 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Johnson, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson PB, Bradley J, Lampotang S, Jackson A, Lizdas D, Johnson W, Brooks E, Vega RBM, Mendenhall N. First-in-human trial using mixed-reality visualization for patient setup during breast or chest wall radiotherapy. Radiat Oncol. 2024 Nov 18;19(1):163. doi: 10.1186/s13014-024-02552-0. PMID 39558366

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Standard of Care, Then HoloLens V2: During treatments 1-5, radiation therapists will position the participant for treatment using the standard of care method.
  During treatments 6-10, radiation therapists will use the hologram the investigators created to initially position the participant for treatment. The participant's final position will be obtained using a standard of care method.
  HoloLens v2: The HoloLens v2 will be used to access the participant's hologram & set the participant up for treatment. Standard of care methods will be utilized to confirm treatment set-up.
- Group 2: HoloLens V2, Then Standard of Care: During treatments 1-5, radiation therapists will use the hologram the investigators created to initially position the participant for treatment. The participant's final position will be obtained using a standard of care method.
  During treatments 6-10, radiation therapists will position the participant for treatment using the standard of care method.
  HoloLens v2: The HoloLens v2 will be used to access the participant's hologram & set the participant up for treatment. Standard of care methods will be utilized to confirm treatment set-up.
Period: First Intervention (Treatments 1-5)
Arm/Group | Group 1: Standard of Care, Then HoloLens V2 | Group 2: HoloLens V2, Then Standard of Care
Started | 13 | 14
Completed | 8 | 12
Not Completed | 5 | 2
Period: Second Intervention (Treatments 6-10)
Arm/Group | Group 1: Standard of Care, Then HoloLens V2 | Group 2: HoloLens V2, Then Standard of Care
Started | 8 | 12
Completed | 8 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Standard of Care, Then HoloLens V2 | Group 2: HoloLens V2, Then Standard of Care | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 4 | 5 | 9
Age, Continuous [Median (Full Range); unit: years] | 53.4 [39.5 to 78.5] | 55.1 [31.2 to 77.7] | 54.9 [31.2 to 78.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Computed Tomography (CBCTs) a Participant Receives During Radiation Therapy Treatment as Quantified Via Counting the Number Used During the Setup Process.
Description: Counting the number of computed tomography a participant receives during radiation therapy treatment as quantified via counting the number used during the setup process
Time Frame: The time frame was from the start of radiation to the 10th fraction of radiation which is approximately two weeks.
Measure: Median (Full Range); unit: number of measurements
Groups:
- Mixed-reality Guided Patient Setup-Group 2 - HoloLens v2 Phase (Treatments 1-5): During treatments 1-5, radiation therapists will use the hologram the investigators created to initially position the participant for treatment. The participant's final position will be obtained using a standard of care method.
  During treatments 6-10, radiation therapists will position the participant for treatment using the standard of care method.
  HoloLens v2: The HoloLens v2 will be used to access the participant's hologram & set the participant up for treatment. Standard of care methods will be utilized to confirm treatment set-up.
Arm/Group | Group 1: Standard of Care, Then HoloLens V2 | Mixed-reality Guided Patient Setup-Group 2 - HoloLens v2 Phase (Treatments 1-5)
Number analyzed (Participants) | 8 | 12
number of measurements
  First Intervention (Treatments 1-5) | 2 [1 to 6] | 3 [1 to 5]
  Second Intervention (Treatments 6-10) | 3 [1 to 7] | 3 [1 to 5]

ADVERSE EVENTS:
Time Frame: Through completion of 7 week radiation therapy course.
Groups:
- Group 1a: Standard of Care (1st Phase); Group 1b: HoloLens V2 (2nd Phase); Group 2b: Standard of Care (2nd Phase): During treatments 1-5, radiation therapists will position the participant for treatment using the standard of care method.
  During treatments 6-10, radiation therapists will use the hologram the investigators created to initially position the participant for treatment. The participant's final position will be obtained using a standard of care method.
  HoloLens v2: The HoloLens v2 will be used to access the participant's hologram & set the participant up for treatment. Standard of care methods will be utilized to confirm treatment set-up.
- Group 2a: HoloLens V2 (1st Phase): During treatments 1-5, radiation therapists will use the hologram the investigators created to initially position the participant for treatment. The participant's final position will be obtained using a standard of care method.
  During treatments 6-10, radiation therapists will position the participant for treatment using the standard of care method.
  HoloLens v2: The HoloLens v2 will be used to access the participant's hologram & set the participant up for treatment. Standard of care methods will be utilized to confirm treatment set-up.
Arm/Group | Group 1a: Standard of Care (1st Phase) | Group 2a: HoloLens V2 (1st Phase) | Group 1b: HoloLens V2 (2nd Phase) | Group 2b: Standard of Care (2nd Phase)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/12 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/12 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 4/8 | 3/12 | 2/8 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1a: Standard of Care (1st Phase) (N=8) | Group 2a: HoloLens V2 (1st Phase) (N=12) | Group 1b: HoloLens V2 (2nd Phase) (N=8) | Group 2b: Standard of Care (2nd Phase) (N=12)
Breast atrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Seroma (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT05178927/Prot_SAP_000.pdf